CLINICAL TRIAL: NCT05353777
Title: Clinical Evaluation of the Levita Robotic Platform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Levita Magnetics (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP007
Record Dates: First submitted 2022-04-12; First posted 2022-04-29 (Actual); Results first posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Bariatric Surgery Candidate; Cholelithiases; Other Disease
MeSH Terms: conditions — Cholelithiasis; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Levita Robotic Platform (Experimental)
  Interventions: Device: Levita Robotic Platform

INTERVENTIONS:
Device: Levita Robotic Platform — Levita Robotic Platform

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of the Levita Robotic Platform (LRP) used with the Levita Magnetic Surgical System (MSS)

DETAILED DESCRIPTION:
Prospective, multi-center, single-arm, open label study designed to assess the safety and feasibility of the use of the Levita Robotic Platform with the Levita Magnetic Surgical System in laparoscopic procedures.

ELIGIBILITY:
Inclusion Criteria:

* • Subject is at least 18 years of age

  * Subject is scheduled to undergo elective laparoscopic procedure
  * Subject signs a written Informed Consent Form (ICF) to participate in the study prior to any study required procedures

Exclusion Criteria:

* • Subjects with pacemakers, defibrillators, or other electromedical implants

  * Subjects with ferromagnetic implants
  * Subjects with significant comorbidities: cardiovascular, neuromuscular, chronic obstructive pulmonary disease, and urological disease (renal failure)
  * Subjects with a clinical history of impaired coagulation confirmed by abnormal blood tests
  * Subject has an anatomical abnormality or disease of intended target tissue noted after initiation of index procedure that would prevent device use
  * Subject is pregnant or wishes to become pregnant during the length of study participation
  * Subject is not likely to comply with the follow-up evaluation schedule
  * Subject is participating in a clinical trial of another investigational drug or device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Robles, MD, Principal Investigator — Hospital FACH
Locations (4):
- Chile (4):
  - Clinica Indisa, Santiago, Santiago Metropolitan
  - Hospital FACH, Santiago, Santiago Metropolitan
  - Hospital San Borja, Santiago, Santiago Metropolitan
  - Hospital Tisne, Santiago, Santiago Metropolitan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Levita Robotic Platform
Started | 48
Completed | 46
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Levita Robotic Platform
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (13.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Chile | 46

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events Related to the Device
Description: Total number of adverse events related to the device.
Time Frame: 30 days
Measure: Number; unit: Adverse events related to device
Arm/Group | Levita Robotic Platform
Number analyzed (Participants) | 46
Adverse events related to device | 3

2. Secondary Outcome: Rate That the Levita Robotic Platform is Able to Engage, Move, and Decouple With the Magnetic Surgical System as Controlled by the Surgeon
Description: Number of successfully performed surgeries without the need of additional tools.
Time Frame: Interoperatively
Measure: Number; unit: Successfully performed surgeries
Arm/Group | Levita Robotic Platform
Number analyzed (Participants) | 46
Successfully performed surgeries | 46

3. Secondary Outcome: Conversion Rate to Open Surgery
Description: Conversion from laparoscopic to open surgery due to inability of the robotic system to provide adequate visualization.
Time Frame: Interoperatively
Measure: Number; unit: Converted procedures
Arm/Group | Levita Robotic Platform
Number analyzed (Participants) | 46
Converted procedures | 0

ADVERSE EVENTS:
Time Frame: Adverse events were documented throughout the course of the study up to thirty (30) days post op.
Arm/Group | Levita Robotic Platform
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 1/46
Other Adverse Events (participants affected / at risk) | 15/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levita Robotic Platform (N=46)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levita Robotic Platform (N=46)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Anal Fissure (Gastrointestinal disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 (3)
Short vessel bleeding (Surgical and medical procedures) | 1 (1)
Nausea and Vomiting (Gastrointestinal disorders) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Liver Capsule Minor Abrasion (Surgical and medical procedures) | 3 (3)
Allergy Rush (Skin and subcutaneous tissue disorders) | 1 (1)
Petechia (Skin and subcutaneous tissue disorders) | 2 (2)
Hematoma (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT05353777/Prot_SAP_000.pdf